CLINICAL TRIAL: NCT03695107
Title: Clinical Study on the Effect of PTH on CYP3A4 Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: XY3-PTH1708A01
Record Dates: First submitted 2018-09-17; First posted 2018-10-03 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- XBDP1-
  Interventions: Drug: Nifedipine controlled released tablets
- XBDP2-
  Interventions: Drug: Nifedipine controlled released tablets

INTERVENTIONS:
Drug: Nifedipine controlled released tablets — lower blood pressure

SUMMARY:
Parathyroid hormone (PTH) may play an important role in the down-regulation of CYP3A4 expression induced by Chronic kidney diseases (CKD). In the study of molecular mechanism, the research group found that the expression of CYP3A2 metabolic enzyme in rat liver decreased in the state of CKD.And PTH may down-regulate the expression of CYP3A4 metabolic enzyme by inhibiting the expression of Nuclear factor- Kilobuse (NF-kB) p65 subunit

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female subjects with an age of 18 or older were included;
* The clinical physician diagnosed CKD with hypertension;
* The physician decided that nifedipine controlled release tablets should be given.
* Subjects agree to the study protocol, clinical and follow-up time, and sign the informed consent after the approval of the ethics committee;
* Subjects will be able to communicate well with the investigator and will be able to complete the study as required.

Exclusion Criteria:

* Patients with CKD requiring dialysis treatment;
* Other clinical reasons that may be considered inappropriate for inclusion by clinicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic renal function associated with hypertension
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-02 (Estimated); Primary Completion 2020-09-10 (Estimated); Study Completion 2020-09-10 (Estimated)

PRIMARY OUTCOMES:
the concentration of nifedipine | at 5-7days
  the concentration of nifedipine

SECONDARY OUTCOMES:
24-hour ambulatory blood pressure | at 1 day and 7day
  mean blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Yang GuoPing, doctor, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University , , China,, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes